CLINICAL TRIAL: NCT00993512
Title: Phase I, Dose-escalating Study to Evaluate Safety and Tolerance of Amphinex Based Photochemical Internalisation (PCI) of Bleomycin in Patients With Local Recurrence or Advanced/Metastatic, Cutaneous or Sub-cutaneous Malignancies
Brief Title: Safety Study of Amphinex Based Photochemical Internalisation (PCI) of Bleomycin in Patients With Cutaneous Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PCI Biotech AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCI 101/06
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Head and Neck Neoplasms; Skin Neoplasms
Keywords: photochemical internalisation; photosensitiser; cutaneous tumour; sub-cutaneous tumour; dose escalation
MeSH Terms: conditions — Head and Neck Neoplasms; Skin Neoplasms | interventions — Bleomycin; Lighting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TPCS2a (Experimental): No comparative treatment is given in this open-label phase I, dose escalating safety study
  Interventions: Drug: Amphinex (TPCS2a); Drug: Bleomycin; Other: Illumination with CeramOptec laser

INTERVENTIONS:
Drug: Amphinex (TPCS2a) — intravenous TPCS2a, followed by standard dose of bleomycin (iv infusion) and illumination with CeramOptec laser.
  Other Names: Amphinex
Drug: Bleomycin — intravenous TPCS2a, followed by standard dose of bleomycin (iv infusion) and illumination with CeramOptec laser.
Other: Illumination with CeramOptec laser — intravenous TPCS2a, followed by standard dose of bleomycin (iv infusion) and illumination with CeramOptec laser.

SUMMARY:
This study is an open, non- randomized, phase I, dose-escalating study to evaluate the safety and tolerance of Amphinex based PCI of bleomycin in patients with local recurrent or advanced/metastatic, cutaneous or sub-cutaneous malignancies.

DETAILED DESCRIPTION:
Eligible patients will be included in cohorts of 3 patients. The initial starting dose for Amphinex will be given 4 days prior to the fixed dose of bleomycin administered by intravenous infusion. The illumination, with red light (laser 652 nm), to the tumour surface and a margin of 2-3 mm outside the tumour surface, will be performed after bleomycin administration.

There will be no comparative procedure in this study. Dose escalation will proceed according to a modification of Simon's accelerated titration design. The number of patients recruited depends on the DLT experienced. A total of 6 patients will be included at each dose level if no more than 1 patient experiences DLT.

Additional cohorts may be added pending the outcome of the previous cohorts and discussions between the investigators and the Sponsor. The primary goal of the study is to assess the safety and tolerance of the Amphinex and determine the maximal tolerated dose (MTD) of Amphinex as a PCI therapy in combination with bleomycin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or above who have given written informed consent.
* Skin type I- IV according to the Fitzpatrick skin classification (see appendix G).
* With a diagnosis of local recurrence or advanced/metastatic, cutaneous or subcutaneous malignancy
* Lesion measurement must not be done more than 2 weeks before the beginning of treatment. More than one field with lesion can be illuminated, but care must be taken to avoid overlap of the fields illuminated.
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, anticancer hormone therapy, or other investigational therapy for at least 2 weeks prior to study entry, and have recovered from the acute effects of therapy.
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Scale (see appendix D).
* Clinically assessed as eligible for bleomycin chemotherapy.
* Have a predicted life expectancy of at least 3 months.
* Geographic proximity that allow adequate follow-up.
* If female: have had childbearing potential either terminated by surgery, radiation, or menopause or attenuated by the use of an approved contraceptive method during and for 3 months after the trial.
* If male: have had reproductive potential either terminated or attenuated by the use of an approved contraceptive method during and for 3 months after the trial.

Exclusion Criteria:

* Have received prior PCI.
* Tumours known to be eroding into a major blood vessel in or adjacent to the illumination site.
* Planned surgery in first 28 days after treatment, except for planned surgical removal of the treated lesion.
* Planned dentist appointments in first 28 days after treatment.
* Anticancer therapy within the first 28 days after treatment.
* Therapy with drugs that induce light sensitivity (e.g. tetracyclines, sulfonamides, phenothiazines, sulfonylurea, hypoglycemic agents, thiazide diuretics, and griseofulvin) within the first 14 days after treatment.
* Co-existing ophthalmic disease likely to require slit-lamp examination within the first 28 days after treatment.
* History of hypersensitivity/anaphylactic reactions.
* Previous cumulative dose of Bleomycin received over 200 000 IE
* Known allergy or sensitivity to photosensitisers.
* Known allergy to Cremophor.
* Known allergy to bleomycin.
* Conditions contraindicated for bleomycin treatment (lung infection, impaired pulmonary function).
* Conditions that worsen when exposed to light (including porphyria).
* Conditions associated with a risk of poor protocol compliance.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 28 days

SECONDARY OUTCOMES:
Tumour response according to Response Evaluation Criteria in Solid Tumors (RECIST) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Colin Hopper, MD, Principal Investigator — University College London Hospitals
Locations (1):
- University College London Hospital, London, United Kingdom

REFERENCES:
- [Derived] Sultan AA, Jerjes W, Berg K, Hogset A, Mosse CA, Hamoudi R, Hamdoon Z, Simeon C, Carnell D, Forster M, Hopper C. Disulfonated tetraphenyl chlorin (TPCS2a)-induced photochemical internalisation of bleomycin in patients with solid malignancies: a phase 1, dose-escalation, first-in-man trial. Lancet Oncol. 2016 Sep;17(9):1217-29. doi: 10.1016/S1470-2045(16)30224-8. Epub 2016 Jul 28. PMID 27475428